CLINICAL TRIAL: NCT00792623
Title: A Phase III, Open-label, Multi-centre Study to Assess the Immunogenicity and Safety of GlaxoSmithKline Biologicals' Live Attenuated Varicella Vaccine (VarilrixTM), Given as a Primary Vaccination at 4.5 Months and 6.5 Months Post-transplantation, in Autologous Stem Cell/ Bone Marrow Transplant Recipients Aged 18 Years and Older.
Brief Title: Immunogenicity and Safety of GSK Biologicals' Live Attenuated Varicella Vaccine (VARILRIXTM).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 208133/178
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2017-04

CONDITIONS: Varicella
Keywords: Varicella; VarilrixTM
MeSH Terms: conditions — Chickenpox

ARMS (1):
- Varilrix Group (Experimental): Subjects with autologous peripheral stem cell/bone marrow transplants, who received 2 doses of Varilrix vaccine subcutaneously in the deltiod region of the non-dominant upper arm, at 4.5 and 6.5 months post-transplantation.
  Interventions: Biological: VarilrixTM

INTERVENTIONS:
Biological: VarilrixTM — Subcutaneous injection, 2 doses, in the deltoid region of the non-dominant upper arm.

SUMMARY:
This study aims to assess the immunogenicity and safety of varicella vaccination in a population of autologous peripheral stem cell/ bone marrow transplantation recipients who have reached at least four months post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

Screening phase:

* A male or female ≥ 18 years of age at the time of study entry.
* Written informed consent obtained from the subject prior to study entry.
* Patients who are planned to undergo autologous peripheral stem cell/ bone marrow transplantation.
* Subjects who the investigator believes can and will comply with the requirements of the protocol
* If the subject is female, she must be of non-childbearing potential; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for 10 months after transplantation.

Active phase:

* Patients who are confirmed to have undergone autologous peripheral stem cell/ bone marrow transplantation.
* If the subject is female, she must be of non-childbearing potential; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for 10 months after transplantation.

Exclusion Criteria:

Screening phase:

* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions in the 10 months post-transplantation.
* History of allergy to any component of the vaccine.
* Patients with difficult to treat disease who are likely to relapse within 6 months post-transplantation.
* Current drug and/or alcohol abuse.

Active phase:

* Use of any investigational or non-registered product (drug or vaccine) during the active phase of the study period.
* Use of immunosuppressants or other immune-modifying drugs within 14 days preceding the administration of the first dose of the study vaccine or planned use during the active phase of the study period.
* Use of rituximab (MabThera) more than 60 days after transplant.
* Administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of vaccine and ending 30 days after.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions in the 10 months post-transplantation.
* History of allergy to any component of the vaccine
* Patients with VZV disease after transplantation and prior to vaccination.
* Ongoing requirement for antiviral therapy with anti-VZV activity beyond 4 months post-transplantation
* Patients with difficult to treat disease who are likely to relapse within 6 months post-transplantation.
* Current drug and/or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-09-08 (Actual); Primary Completion 2007-09-10 (Actual); Study Completion 2007-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Australia (2):
  - GSK Investigational Site, East Melbourne, Victoria
  - GSK Investigational Site, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Sasadeusz J, Prince HM, Schwarer A, Szer J, Stork A, Bock HL, Povey M, Nicholson O, Innis BL. Immunogenicity and safety of a two-dose live attenuated varicella vaccine given to adults following autologous hematopoietic stem cell transplantation. Transpl Infect Dis. 2014 Dec;16(6):1024-31. doi: 10.1111/tid.12295. Epub 2014 Oct 1. PMID 25272081
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 208133/178 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 208133/178 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 208133/178 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 208133/178 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 208133/178 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208133/178 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects in this study were recipients of autologous peripheral stem cell/bone marrow transplants.
Pre-assignment Details: Out of the 45 subjects enrolled in the screening phase of the study, 16 subjects did not receive the study vaccine, as they did not meet eligibility criteria, and were hence eliminated from the study active phase.
Groups:
- Varilrix Group: Subjects with autologous peripheral stem cell/bone marrow transplants, who received 2 doses of Varilrix vaccine subcutaneously in the deltoid region of the non-dominant upper arm, at 4.5 and 6.5 months post-transplantation.
Period: Overall Study
Arm/Group | Varilrix Group
Started | 29
Completed | 22
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Varilrix Group
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.7 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Varicella Vaccine Response
Description: Vaccine response was defined as: for initially seropositive subjects, an antibody titer at Month 8 post-transplantation above or equal to (≥) 4 fold the pre-vaccination antibody titer.
Time Frame: At 8 months post-transplantation = 1.5 months post-second dose of vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity measures and assay results for anti-varicella zoster virus (VZV) antibodies for Month 8 time point were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix Group
Number analyzed (Participants) | 15
Participants | 1

2. Primary Outcome: Anti-varicella Zoster Virus (Anti-VZV) Antibody Titers
Description: Antibody titers were measured by Indirect Immunofluorescence Assay (IFA) and presented as geometric mean titers (GMTs).
Time Frame: At 8 months post-transplantation = 1.5 months post-second dose of vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity measures and assay results for anti-VZV antibodies for Month 8 time point were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Varilrix Group
Number analyzed (Participants) | 15
Titers | 707.5 [308.0 to 1625.5]

3. Secondary Outcome: Number of Subjects With a Varicella Vaccine Response
Description: Vaccine response was defined as: for initially seropositive subjects, antibody titer at 6.5 months post-transplantation ≥ 4 fold the pre-vaccination antibody titer.
Time Frame: At 6.5 months post-transplantation = 2 months post first dose of vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity measures and assay results for anti-VZV antibodies for Month 6.5 time point were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix Group
Number analyzed (Participants) | 10
Participants | 2

4. Secondary Outcome: Number of Seropositive Subjects for Anti-varicella Antibodies
Description: The seropositivity cut-off titer of the assay was an anti-VZV antibody titer greater than or equal to (≥) 1:4.
Time Frame: At pre-transplantation (Month 0), pre-vaccination visit (at 4.5 months post-transplantation), Month 12 and Month 24 (5.5 and 17.5 months post-second dose of vaccination)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects. Only those subjects who provided a serum sample at the specified time point (i.e. with anti-VZV antibody assay results available) were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix Group
Number analyzed (Participants) | 15
Participants
  Month 0 | 15
  Month 4.5 | 15
  Month 12: number analyzed (Participants) | 14
  Month 12 | 14
  Month 24: number analyzed (Participants) | 13
  Month 24 | 13

5. Secondary Outcome: Anti-varicella Antibody Titers
Description: Antibody titers were were measured by Indirect Immunofluorescence Assay (IFA) and presented as geometric mean titers (GMTs).
Time Frame: At pre-transplantation (Month 0), pre-vaccination visit (4.5 months post-transplantation), Month 12 and Month 24 (5.5 and 17.5 post-second dose of vaccination)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Varilrix Group
Number analyzed (Participants) | 15
Titers
  Month 0 | 1024.0 [481.8 to 2176.2]
  Month 4.5 | 645.1 [264.8 to 1571.5]
  Month 12: number analyzed (Participants) | 14
  Month 12 | 380.4 [164.0 to 882.2]
  Month 24: number analyzed (Participants) | 13
  Month 24 | 284.8 [103.8 to 781.5]

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Adverse Events
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 8-day (Days 0-7) post-vaccination period after each dose and across doses
Population: The analysis was performed on the Total vaccinated cohort, which included subjects with at least one vaccination administered. Five subjects who had not completed their symtpom sheets following dose 2 were not included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix Group
Number analyzed (Participants) | 29
Participants
  Any Pain, Dose 1 | 5
  Grade 3 Pain, Dose 1 | 0
  Any Redness, Dose 1 | 4
  Grade 3 Redness, Dose 1 | 0
  Any Swelling, Dose 1 | 0
  Grade 3 Swelling, Dose 1 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 24
  Any Pain, Dose 2 | 4
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 24
  Grade 3 Pain, Dose 2 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 24
  Any Redness, Dose 2 | 3
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 24
  Grade 3 Redness, Dose 2 | 1
  Any Swelling, Dose 2: number analyzed (Participants) | 24
  Any Swelling, Dose 2 | 1
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 24
  Grade 3 Swelling, Dose 2 | 0
  Any Pain, Across Doses | 7
  Grade 3 Pain, Across Doses | 0
  Any Redness, Across Doses | 6
  Grade 3 Redness, Across Doses | 1
  Any Swelling, Across Doses | 1
  Grade 3 Swelling, Across Doses | 0

7. Secondary Outcome: Number of Subjects With Any Fever
Description: Any = fever equal to or greater than (≥) 37.5 °C. Grade 3 fever = fever above (>) 39.0 °C. Related = fever assessed by the investigator as related to the vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period after each dose and across doses
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix Group
Number analyzed (Participants) | 29
Participants
  Any Fever, Dose 1 | 3
  Grade 3 Fever, Dose 1 | 0
  Related Fever, Dose 1 | 0
  Any Fever, Dose 2: number analyzed (Participants) | 24
  Any Fever, Dose 2 | 6
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 24
  Grade 3 Fever, Dose 2 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 24
  Related Fever, Dose 2 | 2
  Any Fever, Across doses | 6
  Grade 3 Fever, Across doses | 0
  Related Fever, Across doses | 2

8. Secondary Outcome: Number of Subjects With Any and Related Rash
Description: Rash was assessed as being either associated to the administration site or not. Non administration site rash was presented by following characteristics (with fever, measles/rubella like, varicella like and related).
Time Frame: During the 43-day (Days 0-42) post-vaccination period after each dose and across doses
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix Group
Number analyzed (Participants) | 29
Participants
  Any Rash, Dose 1 | 3
  Administration site Rash, Dose 1 | 0
  Non-administration site Rash, Dose 1 | 3
  Rash with Fever, Dose 1 | 2
  Measles/Rubella like Rash, Dose 1 | 0
  Varicella like Rash, Dose 1 | 1
  Related non-administration site Rash, Dose 1 | 0
  Any Rash, Dose 2: number analyzed (Participants) | 24
  Any Rash, Dose 2 | 2
  Administration site Rash, Dose 2: number analyzed (Participants) | 24
  Administration site Rash, Dose 2 | 0
  Non-administration site Rash, Dose 2: number analyzed (Participants) | 24
  Non-administration site Rash, Dose 2 | 2
  Rash with Fever, Dose 2: number analyzed (Participants) | 24
  Rash with Fever, Dose 2 | 0
  Measles/Rubella like Rash, Dose 2: number analyzed (Participants) | 24
  Measles/Rubella like Rash, Dose 2 | 0
  Varicella like Rash, Dose 2: number analyzed (Participants) | 24
  Varicella like Rash, Dose 2 | 1
  Related non-administration site Rash, Dose 2: number analyzed (Participants) | 24
  Related non-administration site Rash, Dose 2 | 0
  Any Rash, Across doses | 5
  Administration site Rash, Across Doses | 0
  Non-administration site Rash, Across Doses | 5
  Rash with Fever, Across Doses | 2
  Measles/Rubella like Rash, Across doses | 0
  Varicella like Rash, Across doses | 2
  Related non-administration site Rash, Across doses | 0

9. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period after each dose and across doses
Population: The analysis was performed on the Total vaccinated cohort, which included subjects with at least one vaccination administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix Group
Number analyzed (Participants) | 29
Participants | 11

10. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the active phase of the study (up to Month 24)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix Group
Number analyzed (Participants) | 29
Participants | 5

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 8-day (Days 0-7) post-vaccination period; Unsolicited AEs: during the 43-day (Days 0-42) post-vaccination period; Serious adverse events (SAEs): during the entire study, up to Month 24 post-transplantation.
Arm/Group | Varilrix Group
All-Cause Mortality (participants affected / at risk) | 1/29
Serious Adverse Events (participants affected / at risk) | 5/29
Other Adverse Events (participants affected / at risk) | 14/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varilrix Group (N=29)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varilrix Group (N=29)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 6 (7)
Injection site pruritus (General disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Pain (General disorders) | 7 (9)
Upper respiratory tract infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.